CLINICAL TRIAL: NCT05007548
Title: An Open-label, Comparative Phase II Clinical Trial to Assess the Accuracy and Reliability of the Ga68-Dolacga Positron Emission Tomography Compared to Computer Tomography Volumetry and Indocyanine Green Retention Test for Measurement of Liver Reserve Among Scheduled Surgery Operation Patients
Brief Title: to Assess the Accuracy and Reliability of the Ga68-Dolacga Positron Emission Tomography Compared to Computer Tomography Volumetry and Indocyanine Green Retention Test for Measurement of Liver Reserve
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Atomic Research Institute, Taiwan (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: INER-V09DX-02
Record Dates: First submitted 2021-07-29; First posted 2021-08-16 (Actual); Last update posted 2023-12-13 (Actual); Status verified 2023-12

CONDITIONS: Hepatic Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Ga68-Dolacga Injection (Experimental): Ga68-Dolacga will be administered via iv bolus injection followed by a whole-body PET/CT scan for liver reserve evaluation.
  Interventions: Drug: Ga68-Dolacga Injection

INTERVENTIONS:
Drug: Ga68-Dolacga Injection — Ga68-Dolacga Injection, 2.0±1.0 mCi, single dose, iv bolus
  Other Names: Ga68-INER038

SUMMARY:
This is a phase 2 open-labeled study to compare the Ga68-Dolacga positron emission tomography with computer tomography volumetry and indocyanine green retention test for measurement of liver reserve among scheduled surgery operation patients.

DETAILED DESCRIPTION:
This is a phase 2 open-labeled study to compare the Ga68-Dolacga positron emission tomography with computer tomography volumetry (CTV) and indocyanine green retention test (ICGR15) for measurement of liver reserve among scheduled surgery operation patients. The goal is to enroll 30 eligible subjects scheduled for surgery operation.

CTV and ICGR15 will occur within 7 days prior to the imaging visit for all eligible subjects. During the imaging visit (visit 2, Day 1), subjects will receive an iv bolus injection of 2.0±1.0 mCi Ga68-Dolacga Injection. Ga68-Dolacga PET will be kinetically performed 60 minutes immediately after iv injection.

Two follow-up visits (visit 3 at Day 7±2 and visit 4 at Day 14±2) will be conducted to confirm subject well-being and to collect information about any new adverse events (if any).

ELIGIBILITY:
Inclusion Criteria:

1. Scheduled operation subjects with diagnosed hepatic carcinoma. The eligibility criteria for operation refer to protocol Appendix II: Diagnosis and Treatment Guidelines for Hepatocellular Carcinoma in Chang Gung Memorial Hospital;
2. Subjects without ascites or with controllable ascites;
3. Serum total bilirubin level < 2.0 mg/dL;
4. Written informed consent must be obtained before any assessment is performed.
5. Male or female subjects aged 20 or above, inclusive, at date of consent.

Exclusion Criteria:

1. Presence of distant metastases;
2. A body weight loss of >10% during the 6 months before operation;
3. Presence of seriously impaired function of vital organs due to respiratory, renal, or heart disease;
4. Cholangiocarcinoma;
5. General PET exclusion criteria;
6. Pregnant women, lactating or breast-feeding women;
7. Patient who can't be followed up for any reason.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2021-12-14 (Actual); Primary Completion 2023-11-20 (Actual); Study Completion 2023-11-20 (Actual)

PRIMARY OUTCOMES:
Measurement of liver reserve obtained from Ga68-Dolacga PET performed in patients scheduled surgical operation (Percentage of injection dose, %ID) | visit 2 (Day 1)
  The liver reserve obtained from Ga68-Dolacga PET is expressed in "percentage of injection dose (%ID)."
Measurement of liver reserve obtained from CTV performed in patients scheduled surgical operation (Remnant volume rate (%)) | within 7 days prior to Day 1
  The liver reserve obtained from computer tomography volumetry (CTV) is expressed in "remnant volume rate (%)."
Measurement of future liver remnant volume rate (FLRV%) | within 7 days prior to Day 1
  The future liver remnant volume rate (FLRV%) is calculated by dividing the future remnant liver volume by the total functional liver volume from CTV and expressed as %.
Measurement of future liver remnant function rate (FLRF%) | visit 2 (Day 1)
  The future liver remnant function rate (FLRV%) is calculated by dividing the uptake in the future remnant liver volume by the uptake in the total liver volume from Ga68-Dolacga PET and expressed as %.
Correlation of the percentage of injection dose (%ID) in liver determined by Ga68-Dolacga PET with conventional liver function tests | from pre-dose to Day 1
  The conventional liver function tests parameters include alanine aminotransferase (U/L), aspartate aminotransferase (U/L), total bilirubin (mg/dL), direct bilirubin (mg/dL), gamma-glutamyl transpeptidase (U/L), total protein (g/dL), albumin/globulin ratio, albumin (g/dL), prothrombin time/International Normalized Ratio (PT/INR), platelet count (×10^3/μL), ICGR15 (%), Child-Pugh classification (Class A to Class C), MELD score.
Correlation of the remnant volume rate determined by CTV with conventional liver function tests | from pre-dose to Day 1
  The conventional liver function tests parameters include alanine aminotransferase (U/L), aspartate aminotransferase (U/L), total bilirubin (mg/dL), direct bilirubin (mg/dL), gamma-glutamyl transpeptidase (U/L), total protein (g/dL), albumin/globulin ratio, albumin (g/dL), prothrombin time/International Normalized Ratio (PT/INR), platelet count (×10^3/μL), ICGR15 (%), Child-Pugh classification (Class A to Class C), MELD score.
Correlation of the ICGR15 with the conventional liver function tests | from pre-dose to Day 1
  The conventional liver function tests parameters include alanine aminotransferase (U/L), aspartate aminotransferase (U/L), total bilirubin (mg/dL), direct bilirubin (mg/dL), gamma-glutamyl transpeptidase (U/L), total protein (g/dL), albumin/globulin ratio, albumin (g/dL), prothrombin time/International Normalized Ratio (PT/INR), platelet count (×10^3/μL), Child-Pugh classification (Class A to Class C), MELD score.

SECONDARY OUTCOMES:
Correlation of the percentage of injection dose (%ID) in liver determined by Ga68-Dolacga PET with the fibrosis indices | from pre-dose to Day 1
  The fibrosis indices include liver stiffness measurement (kPa) determined by Fibroscan and the Fibrosis-4 (FIB-4) index.
Correlation of the ICGR15 with the fibrosis indices | from pre-dose to Day 1
  The fibrosis indices include liver stiffness measurement (kPa) determined by Fibroscan and the Fibrosis-4 (FIB-4) index.
Number of subjects with clinically significant changes in systolic blood pressure and diastolic blood pressure | from pre-dose to 14±2 days post dose
Number of subjects with body temperature abnormalities | from pre-dose to 14±2 days post dose
Number of subjects with clinically significant changes in Heart Rate | from pre-dose to 14±2 days post dose
Number of subjects reporting clinically significant changes in serum biochemical tests | from pre-dose to 14±2 days post dose
Number of subjects reporting clinically significant changes in hematological tests | from pre-dose to 14±2 days post dose
Number of subjects reporting clinically significant changes in urinalysis | from pre-dose to 14±2 days post dose
Number of subjects with clinically significant changes in electrocardiogram(ECG) | from pre-dose to 14±2 days post dose
  The ECG parameters include: PR interval (milliseconds), QTc interval (milliseconds), QRS duration (milliseconds)
Incidence of Adverse Events (AEs) and Serious Adverse Events (SAEs) | 14 days
  All laboratory abnormalities which are compared with screening values and out of the reference range will be considered as AE and will be assessed its relationship to the study drug. Any ECG changes including ECG waveform will be assessed as AE(s) and will be followed to assess whether they resolved and when they resolved.
Incidence of posthepatectomy liver failure (PHLF) | on or after postoperative day 5 (POD 5)
Severity grading of PHLF as defined by the International Study Group of Liver Surgery (ISGLS) | on or after postoperative day 5 (POD 5)
  Subjects diagnosed with PHLF are classified as grade A, grade B or grade C based on its severity.
Comparison of CTV and Ga68-Dolacga PET parameters in patients with PHLF | on or after postoperative day 5 (POD 5)
  Following parameters will be compared:
  * liver reserve obtained from CTV vs liver reserve obtained from Ga68-Dolacga PET
  * FLRV% vs FLRF%

CONTACTS AND LOCATIONS:
Overall Officials: Wei-Chen Lee, MD, Principal Investigator — Linkon Chang Gung Memorial Hospital
Locations (1):
- Linkon Chang Gung Memorial Hospital, Taoyuan, Taiwan

IPD SHARING:
Plan to Share IPD: No